CLINICAL TRIAL: NCT00002174
Title: Further Evaluation of Thalidomide's Ability to Potentiate the Immune Response to HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 262A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections
Keywords: Adjuvants, Immunologic; Thalidomide; Cytokines; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
To determine if Thalidomide modulates the production of HIV-suppressor factors (MIP-1 alpha, MIP-1 beta, Rantes) and TH1 type cytokines (IL-12 and INF-gamma) in HIV-infected patients and alters viral load.

DETAILED DESCRIPTION:
Patients will be divided, 5 per group, into Groups I, II, III and IV. Groups I and II will include patients who have decided not to take anti-retro viral drugs. Groups III and IV will include patients receiving the same types of antiretroviral drugs. Patients in groups I and III will receive thalidomide while patients in group II and IV will receive placebo. The placebo capsules will be the same color as the thalidomide capsules and will contain glucose powder. Patients will ingest one capsule of thalidomide at 9 PM daily on days 0, 1, 2, 3, 4, 5 and 6.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4+ cell count >= 200/microliter or > 14% CD4+ cells in peripheral blood.
* Willingness to commit to the study duration and agree to abide to the time table for entry into the study, ingestion of thalidomide and follow-up.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions or symptoms are excluded:

* Fertile females.
* Patients who participated in a clinical study involving a new drug or device within the last 2 months or the period of time equivalent to seven times the half life of the study drug, whichever is longer.

Patients with any of the following prior conditions are excluded:

HIV related pre-existing peripheral neuropathy.

Prior Medication:

Excluded:

Patients using systemic steroidal anti inflammatory drugs or pentoxifylline within 10 days of dosing with thalidomide.

Required:

10 of the 20 patients must be on antiretroviral therapy and the other 10 will be subjects who have decided not to be on any antiretroviral drug prior to enrollment into this study and do not plan to start such treatment during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Clinic, New Orleans, Louisiana, United States